CLINICAL TRIAL: NCT02491177
Title: Maximizing Adherence and Retention for Women and Infants in the Context of Option B+
Brief Title: Mother and Infant Visit Adherence and Treatment Engagement Study
Acronym: MOTIVATE!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Alabama at Birmingham (Other); Kenya Medical Research Institute (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 14-0331; R01HD080477-01 (NIH)
Record Dates: First submitted 2015-03-11; First posted 2015-07-07 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV Transmission; Prevention of Mother to Child Transmission; Linkage to care; Retention in care; Community Mentor Mothers; Mobile phone text messaging; Antiretroviral therapy adherence; Infant Health; Maternal CD4/viral loads; Early infant diagnosis; Acceptability of interventions; Vertical transmission
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- cMM and Text Messaging (Other): Participants randomized to this arm will receive both the community mentor mother and mobile phone text messaging intervention. The community mentor mother intervention will consist of home visits conducted by the community mentor mother who will assist with safe disclosure, support safe infant feeding, promote safer sex and family planning, encourage early infant testing and follow up, and promote ART adherence and return for HIV care visits. The text messaging intervention will entail participants receiving tailored mobile phone text messages at their preferred frequency and in their preferred language.
  Interventions: Behavioral: cMM; Behavioral: Text Messaging
- cMM Only (Other): Participants randomized to this arm will receive the community mentor mother intervention only.The community mentor mother intervention will consist of home visits conducted by the community mentor mother who will assist with safe disclosure, support safe infant feeding, promote safer sex and family planning, encourage early infant testing and follow up, and promote ART adherence and return for HIV care visits.
  Interventions: Behavioral: cMM
- Text Messaging Only (Other): Participants randomized to this arm will receive the mobile phone text messaging intervention only. The text messaging intervention will entail participants receiving tailored mobile phone text messages at their preferred frequency and in their preferred language.
  Interventions: Behavioral: Text Messaging
- Neither cMM nor Text Messaging (No Intervention): Participants randomized to this arm will receive standard of care with no interventions.

INTERVENTIONS:
Behavioral: cMM — Home visits from community mentor mothers
  Arms: cMM Only; cMM and Text Messaging
Behavioral: Text Messaging — Text messages received on mobile phone
  Arms: Text Messaging Only; cMM and Text Messaging

SUMMARY:
This is a 2x2 factorial cluster randomized trial of two interventions to improve retention and adherence for women and infants on Option B+. The overall goal is to determine which intervention (or combination of interventions) maximizes antiretroviral therapy (ART) adherence and retention in care in the context of Option B+ and thus improves maternal and infant health outcomes.The proposed study will be conducted in rural Nyanza Province, Kenya at 20 low-resource primary health care facilities and associated communities supported by Family AIDS Care and Education Services (FACES), a President's Emergency Plan for AIDS Relief (PEPFAR)-funded HIV prevention care, and treatment program, ((AIDS) acquired immune deficiency syndrome, (HIV) human immunodeficiency virus) . The investigators will assess both process and outcome indicators using a 2x2 factorial design, in which equal numbers of clusters will be randomized to one of the interventions (community-based mentor mothers or theory-based mobile text messages), both interventions, or standard of care. The interventions will be added to fully integrated high quality HIV and antenatal, maternal, neonatal, and child health (ANC/MNCH) services already offered at these sites.

DETAILED DESCRIPTION:
In order to eliminate new pediatric HIV infections, save maternal lives, and simplify antiretroviral therapy (ART) implementation in settings with generalized HIV epidemics, current World Health Organization (WHO) guidance recommends lifelong triple ART for all pregnant and breastfeeding women (Option B+). However, despite the promise of Option B+ to remove logistical barriers and to promote maternal health through life-long ART, this strategy brings challenges. Key amongst these challenges are adherence to ART and continuous retention in HIV care, especially for women who do not require ART for their own health. Barriers to adherence and retention in care for prevention of mother-to-child transmission (PMTCT) have been identified at the individual, interpersonal, community, and health facility levels; yet specific barriers in the context of Option B+ are not well understood. The investigators' study will be conducted at 20 health facilities and associated communities in Nyanza Province, Kenya where Mother to Child Transmission (MTCT) rates prior to Option B+ roll-out remained near 10%, despite the wide availability of PMTCT services. As Option B+ is scaled up in Kenya, it is essential to identify effective methods to ensure long-term adherence and retention in care for mother-baby pairs, throughout pregnancy, breastfeeding, and beyond. Building on the investigating team's prior research experience in this setting, the investigators propose to gain understanding of and address potential barriers at the individual, community, and health facility levels through formative research with HIV-positive pregnant and postpartum women, their male partners, and health care providers. This information will be used to refine two proposed interventions that are highly likely to maximize ART adherence and retention in care among HIV-infected pregnant women and HIV-exposed infants. These interventions will be rigorously tested in rural Kenya, using a cluster randomized 2x2 factorial design. The evidence-based interventions to be tested will include 1) community Mentor Mothers (cMM) who will provide support for ART adherence and retention in care for HIV-positive women in the community and 2) individually tailored, theory based mobile phone text messages to help retain women and infants in HIV care. The investigators' overall goal is to determine which intervention (or combination of interventions) maximizes ART adherence and retention in care in the context of Option B+ and thus improves maternal and infant health outcomes. The investigators' primary outcomes will include ART adherence at 12 months postpartum and retention in care, measured by a documented HIV care visit within 90 days prior to 12 months postpartum. Secondary outcomes will include MTCT at 6 weeks, 12 months and 18 months; as well as maternal viral loads and CD4 counts. Results from this study will inform the scale-up of Option B+ in Kenya by identifying effective interventions and combinations of interventions that can reduce barriers and increase facilitators of optimal ART adherence and retention in care with the aims of reaching the elimination of mother to child transmission of HIV and significantly improving maternal health.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older,
* HIV-infected pregnant women and their HIV-exposed infants pairs,
* attends the antenatal care (ANC) clinic at one of the study sites.

Exclusion Criteria:

* Less than 18 years of age,
* HIV-infected women not currently pregnant,
* not HIV-infected at the time of the first ANC visit.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1338 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Self-reported adherence on antiretroviral therapy | 12 months post-partum
  Self-report
Adherence on antiretroviral therapy | 12 months post-partum
  Viral load<100 copies/ml based on medical records
Adherence on antiretroviral therapy (infant) | 12 months post-partum
  Use of ARVs for the infant
Retention in care | 12 months post-partum
  Proportion of women who have an HIV care visit within 90 days at 12 months after the birth
Adherence on antiretroviral therapy (dried blood spots) | 12 months post-partum
  Viral load<100 copies/ml based on dried blood spots

SECONDARY OUTCOMES:
Maternal CD4 count change | 6 months after baseline
  Change in CD4 count baseline to 6 months after baseline
Maternal viral load count change | 6 months after baseline
  Change in viral load from baseline to 6 months after baseline
Infant retention in care (feeding method) | 12 and 18 months
  Infant feeding method
Infant retention in care | 12 and 18 months
  Retention in care through 12 and 18 months
Infant retention in care (survival status) | 12 and 18 months
  Survival status of infant
Uptake of intervention services (Number/types of text messages sent) | 3 years
  Number/types of text messages sent
Uptake of intervention services (receipt of text messages) | 3 years
  Receipt of text messages
Uptake of intervention services (home visits) | 3 years
  Number of home visits received
Uptake of intervention services (support groups attended) | 3 years
  Number of support groups attended.
Mother-to-Child-Transmission | 6 weeks, 9 months and 18 months
  Result of infant HIV test at 6 wks, 9,18 months
Infant testing | 6 weeks, 9 months and 18 months
  Uptake and date of infant testing
Infant enrollment in care | 6 weeks
  Infant enrollment in HIV care
Male partner involvement | 12 months post-partum
  Composite variable including Y/N response to indicate if male partner attended a health visit with his female partner, encouraged facility delivery, reminded to take HIV medication, reminded to go for HIV care, provided transport money to go to the clinic/dispensary, reminded to give the infant prophylaxis, helped giving the infant prophylaxis medication, collected medication for the woman or infant, encouraged specific infant feeding, and encouraged pediatric HIV testing. These are assessed in the follow-up questionnaires completed at 12 months post-partum.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Abuogi, MD, MSc, Principal Investigator — University of Colorado, Denver
Locations (1):
- Kenya Medical Research Institute, Nairobi, Kenya

REFERENCES:
- [Derived] Abuogi LL, Onono M, Odeny TA, Owuor K, Helova A, Hampanda K, Odwar T, Onyango D, McClure LA, Bukusi EA, Turan JM. Effects of behavioural interventions on postpartum retention and adherence among women with HIV on lifelong ART: the results of a cluster randomized trial in Kenya (the MOTIVATE trial). J Int AIDS Soc. 2022 Jan;25(1):e25852. doi: 10.1002/jia2.25852. PMID 35041776
- [Derived] Helova A, Onono M, Abuogi LL, Hampanda K, Owuor K, Odwar T, Krishna S, Odhiambo G, Odeny T, Turan JM. Experiences, perceptions and potential impact of community-based mentor mothers supporting pregnant and postpartum women with HIV in Kenya: a mixed-methods study. J Int AIDS Soc. 2021 Nov;24(11):e25843. doi: 10.1002/jia2.25843. PMID 34797955
- [Derived] Onono M, Odwar T, Wahome S, Helova A, Bukusi EA, Hampanda K, Turan J, Abuogi L. Behavioral Interventions can Mitigate Adverse Pregnancy Outcomes Among Women Conceiving on ART and Those Initiated on ART During Pregnancy: Findings From the MOTIVATE Trial in Southwestern Kenya. J Acquir Immune Defic Syndr. 2021 Jan 1;86(1):46-55. doi: 10.1097/QAI.0000000000002521. PMID 33306563
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276
- [Derived] Wanga I, Helova A, Abuogi LL, Bukusi EA, Nalwa W, Akama E, Odeny TA, Turan JM, Onono M. Acceptability of community-based mentor mothers to support HIV-positive pregnant women on antiretroviral treatment in western Kenya: a qualitative study. BMC Pregnancy Childbirth. 2019 Aug 13;19(1):288. doi: 10.1186/s12884-019-2419-z. PMID 31409297
- [Derived] Odeny TA, Onono M, Owuor K, Helova A, Wanga I, Bukusi EA, Turan JM, Abuogi LL. Maximizing adherence and retention for women living with HIV and their infants in Kenya (MOTIVATE! study): study protocol for a randomized controlled trial. Trials. 2018 Jan 29;19(1):77. doi: 10.1186/s13063-018-2464-3. PMID 29378622